CLINICAL TRIAL: NCT06064240
Title: Evaluation of Changes in Liver Fat Content and Exploration of Potential Effect Actors After Bariatric Surgery Based on MRI
Brief Title: Liver Fat Content and Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: yu li，MD (Other)
Responsible Party: Sponsor-Investigator, yu li，MD, Doctoral, The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Other Study IDs: liyu
Record Dates: First submitted 2023-09-21; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Bariatric Surgery; Magnetic Resonance Imaging
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Before operation, 1 month after operation, 3 months after operation and 6 months after operation.: Patients who underwent bariatric surgery were followed up regularly before and after surgery.
  Interventions: Other: We do not have any intervention type

INTERVENTIONS:
Other: We do not have any intervention type — We do not have any intervention type

SUMMARY:
On the basis of previous research, this subject intends to evaluate the liver improvement of patients with liver disease after weight loss by MRI, and quantify it by extracting features, so as to provide a new method to judge the liver status of patients with liver disease, and to evaluate the correlation between the inflammatory status of patients and the quantitative features of MRI, and try to explain the reasons for the improvement of fatty liver status of patients with liver disease after weight loss. To provide a new theoretical basis for fatty liver and systemic inflammatory liver damage in patients with liver disease after weight loss surgery, and to link them, and try to explain the improvement of fatty liver in patients with liver disease through the reduction of systemic inflammatory level.

DETAILED DESCRIPTION:
This study is a prospective study to explore the improvement of fatty liver and severe state of the whole body in patients with liver disease undergoing weight-loss surgery. The research object is obese patients who underwent laparoscopic sleeve gastrectomy in our hospital. According to the standard of accepting the discharge, about 50 patients were selected and divided into groups according to preoperative, postoperative one month, postoperative three months and postoperative six months.All patients underwent routine sequence examinations using a Siemens 3.0T MRI scanner (MAGNETOM Prisma, Siemens Healthcare, Munich, Germany).This study investigates alterations in NAFLD among patients with obesity who underwent bariatric surgery using MRI-PDFF and MRS techniques. Additionally, we evaluated the factors that may influence these changes in patients after the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* 16 years old < age < 60 years old
* BMI > 32kg/m2
* No previous drinking history; weekly drinking of males < 210g and females < 140g in 12 months
* Preoperative auxiliary examination supports the diagnosis of fatty liver, and liver MRI examination
* Previous attempts to lose weight are ineffective
* Complete case data.

Exclusion criteria:

* Secondary obesity
* History of drinking or excessive drinking (in the past 12 months, male's weekly alcohol intake was ≥210g, female's weekly alcohol intake was ≥ 140g)
* Other diseases causing abnormal liver function
* Body mass index < 28kg/m2
* Poor compliance or self-control, unable to follow the dietary guidance after operation
* Those who cannot complete the follow-up

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The major Study Population were who had accept the bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Liver fat fraction | before surgery、one 、three、six month after surgery
  The primary outcome was a indicator for evaluating liver fat content.
white blood cell | before surgery、one 、three、six month after surgery
  The primary outcome was a indicator for evaluating inflammation.
aspartate aminotransferase | before surgery、one 、three、six month after surgery
  The primary outcome was a indicator for evaluating liver function.
alanine aminotransferase | before surgery、one 、three、six month after surgery
  The primary outcome was a indicator for evaluating liver function.
C-reactive protein | before surgery、one 、three、six month after surgery
  The primary outcome was a indicators for evaluating inflammation.
neutrophile granulocyte | before surgery、one 、three、six month after surgery
  The primary outcome was a indicator for evaluating inflammation.

SECONDARY OUTCOMES:
low-density lipoprotein | before surgery、one 、three、six month after surgery
  The secondary outcome was a indicator for evaluating blood fat.
high-density lipoprotein | before surgery、one 、three、six month after surgery
  The secondary outcome was a indicator for evaluating blood lipid.
glucose | before surgery、one 、three、six month after surgery
  The secondary outcome was a indicator for evaluating blood glucose.

OTHER OUTCOMES:
Body Mass Index | before surgery、one 、three、six month after surgery
  The pre-specified outcome was a indicator for evaluating effectiveness of bariatric surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao University Affiliated Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No